CLINICAL TRIAL: NCT06357455
Title: Platelet Count and Function After Usage of Two Different Cell Saver Devices During Liver Transplant Surgery: A Randomized Controlled Bi-Center Equivalence Trial
Brief Title: Platelet Count and Function After Usage of Two Different Cell Saver Devices During Liver Transplant Surgery
Acronym: PLFLTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eduardo Schiffer (Other)
Collaborators: University Hospital, Geneva (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor-Investigator, Eduardo Schiffer, Professor, Head of Unit, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Platelet CellSaver Liver trnsp
Record Dates: First submitted 2024-03-26; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Liver Transplant; Hemorrhage, Surgical
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAME™ Device group (Experimental): SAME™ Autotransfusion Device that is being tested for recovery of platelets along with RBCs
  Interventions: Device: Cell Salvage Autotransfusion: SAME™ device
- Autolog™ Device group (Active Comparator): Autolog™ standard autotransfusion device currently used at our institution
  Interventions: Device: Cell Salvage Autotransfusion: Autolog™ device

INTERVENTIONS:
Device: Cell Salvage Autotransfusion: SAME™ device — * Intervention studied: processing of salvaged blood using the SAME™ autotransfusion device
  * Population studied: 20 patients planned to undergo high-risk liver transplantation.
  * "Treatment" group.
  All perioperative measures will be performed according to international, national and in-house standards.
  Arms: SAME™ Device group
Device: Cell Salvage Autotransfusion: Autolog™ device — * Intervention studied: processing of salvaged blood using the Autolog™ (Medtronic) autotransfusion device (in-house standard device).
  * Population studied: 20 patients planned to undergo high-risk liver transplantation.
  * "Control" group
  All perioperative measures will be performed according to international, national and in-house standards.
  Arms: Autolog™ Device group

SUMMARY:
Intraoperative cell salvage is commonly used in surgeries that carry a major hemorrhagic risk to reduce the administration of allogeneic red blood cells and thus improve the outcome for the patient. When processing the salvaged blood, however, a large part of the patient's plasma is washed out. This is a disadvantage with regard to an optimal coagulation status after these types of surgeries, especially liver transplantation.

There are currently various cell saver systems on the market. According to the manufacturers, the plasma is returned to the patient in different quantities as part of the processing procedure. Thus, it can be assumed that in addition to red blood cells, platelets (part of plasma) are re-transfused and contribute to an optimized coagulation. Unfortunately, there is a lack of studies in this regard in the liver transplant surgery population.

The investigators aim to study the performance of two different cell saver devices regarding preservation of platelet number and function.

DETAILED DESCRIPTION:
- Study design: Randomized controlled bi-center trial

* Primary objective: to compare platelet number and function after processing and re-transfusion of the salvaged blood to the patient by using different cell saver devices.
* Secondary (main) objectives: to compare a) the coagulation profile and b) the usage of blood products (frequency of administration of labile and stable blood products).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing liver transplantation surgery

Exclusion Criteria:

* Age < 18 years old
* Active liver malignancy
* Preoperative use of oral or intravenous anti-coagulants or antiplatelet agents (except aspirin)
* Inability to understand and sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Platelet number | Day 1
  Platelet number will be measured using flow cytometry in the laboratory after processing and after retransfusion of the salvaged blood to the patient.

SECONDARY OUTCOMES:
Platelet function | Day 1
  Platelets function will be assessed by multiple electrode aggregometry (Multiplate® analyzer, Roche Diagnostics, Mannheim, Germany).
Platelet function | Day 1
  Platelets function will be measured by platelet activation markers (P-selectin)
Platelet function | Day 1
  Platelets function will be measured by platelet activation markers (GPIb)
Platelet function | Day 1
  Platelets function will be measured by platelet activation markers (GPIIb)
Platelet function | Day 1
  Platelets function will be measured by point-of-care test (ClotPro, Hemonetics Corporation, Boston, MA, USA) using ExTest.
Platelet function | Day 1
  Platelets function will be measured by point-of-care test (ClotPro, Hemonetics Corporation, Boston, MA, USA) using FibTest assays.
Blood plasma albumin level | Day 1
  measured by spectrophotometry
Blood hemoglobin level | Day 1
  measured by spectrophotometry
Blood lactate level | Day 1
  measured by spectrophotometry
Free hemoglobin level | Day 1
  measured by spectrophotometry
Anti-Xa activity | Day 1
  measured by Anti-Xa assay
Number of allogeneic blood products used | Day 1
  Number of allogeneic blood products used (red blood cell, fresh frozen plasma, platelet concentrates) until ICU discharge
Number of coagulation concentrates used | Day 1
  Number of coagulation concentrates used (prothrombin complex concentrate, fibrinogen concentrate) until ICU discharge
Amount of autologous blood at the end of the liver transplantation | Day 1
  Amount of autologous blood at the end of the liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Schiffer, MD, Study Director — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Background] Mansour A, Beurton A, Godier A, Rozec B, Zlotnik D, Nedelec F, Gaussem P, Fiore M, Boissier E, Nesseler N, Ouattara A. Combined Platelet and Red Blood Cell Recovery during On-pump Cardiac Surgery Using same by i-SEP Autotransfusion Device: A First-in-human Noncomparative Study (i-TRANSEP Study). Anesthesiology. 2023 Sep 1;139(3):287-297. doi: 10.1097/ALN.0000000000004642. PMID 37294939
- [Background] Mansour A, Decouture B, Roussel M, Lefevre C, Skreko L, Picard V, Ouattara A, Bachelot-Loza C, Gaussem P, Nesseler N, Gouin-Thibault I. Combined Platelet and Erythrocyte Salvage: Evaluation of a New Filtration-based Autotransfusion Device. Anesthesiology. 2021 Aug 1;135(2):246-257. doi: 10.1097/ALN.0000000000003820. PMID 33984126
- [Background] Klein AA, Bailey CR, Charlton AJ, Evans E, Guckian-Fisher M, McCrossan R, Nimmo AF, Payne S, Shreeve K, Smith J, Torella F. Association of Anaesthetists guidelines: cell salvage for peri-operative blood conservation 2018. Anaesthesia. 2018 Sep;73(9):1141-1150. doi: 10.1111/anae.14331. Epub 2018 Jul 10. PMID 29989144
- [Background] Sikorski RA, Rizkalla NA, Yang WW, Frank SM. Autologous blood salvage in the era of patient blood management. Vox Sang. 2017 Aug;112(6):499-510. doi: 10.1111/vox.12527. Epub 2017 Jun 5. PMID 28580663
- [Background] Schreiber K, Decouture B, Lafragette A, Chollet S, Bruneau M, Nicollet M, Wittmann C, Gadrat F, Mansour A, Forest-Villegas P, Gauthier O, Touzot-Jourde G. A novel autotransfusion device saving erythrocytes and platelets used in a 72 h survival swine model of surgically induced controlled blood loss. PLoS One. 2022 Mar 24;17(3):e0260855. doi: 10.1371/journal.pone.0260855. eCollection 2022. PMID 35324911